CLINICAL TRIAL: NCT07204106
Title: Efficacy of Dexmedetomidine Nasal Spray Combined With Propofol for Deep Sedation in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP): A Prospective Randomized Study
Brief Title: Efficacy Study of Dexmedetomidine Nasal Spray Combined With Propofol for Deep Sedation in ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiyou Wei (Other)
Collaborators: Shanghai East Hospital of Tongji University (Other)
Responsible Party: Sponsor-Investigator, Shiyou Wei, Department of Anesthesiology, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250527IIT0060
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Dexmedetomidine Induced Sedation; Nasal Administration; Sprays
Keywords: Dexmedetomidine; Nasal Spray; Sedation; ERCP
MeSH Terms: interventions — Dexmedetomidine; Nasal Sprays; Propofol; Sufentanil; Saline Solution

STUDY DESIGN:
Intervention Model Description: Three-group, parallel-controlled trial, designed to investigate the efficacy and safety of dexmedetomidine nasal spray in the application of ERCP (Endoscopic Retrograde Cholangiopancreatography), serving as a substitute for intravenous pump infusion of dexmedetomidine.
Who Masked: Participant
Masking Description: While the anesthesiologists who collected data during ERCP were not blinded, they were excluded from analyzing the follow-up results. The anesthesia was administered by the same experienced anesthesiologist, with post-anesthesia evaluation and follow-up care handled by a different physician. Neither the patients nor the data collectors were aware of the sedation protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group ① (Experimental): Dexmedetomidine Nasal Spray Group
  Interventions: Drug: Dexmedetomidine Injection (nasal spray) + Propofol Injection + Sufentanil Injection
- Experimental Group ② (Active Comparator): Dexmedetomidine Intravenous Group
  Interventions: Drug: Normal Saline (nasal spray) + Dexmedetomidine Injection (intravenous) + Propofol Injection + Sufentanil Injection
- Control Group (Sham Comparator): Propofol Alone Group
  Interventions: Drug: Regular sedation protocol

INTERVENTIONS:
Drug: Dexmedetomidine Injection (nasal spray) + Propofol Injection + Sufentanil Injection — 1. Preoperative intervention：30 minutes before entering the operating room, 50-100μg of Dexmedetomidine Injection is administered via nasal spray in the anesthesia preparation room.
  2. Induction phase：Intravenous injection of Sufentanil Injection (Yichang Renfu Pharmaceutical Co., Ltd.) at a dose of 0.1μg/kg, and Propofol Injection (Jiabo Pharmaceutical, Guangdong, China) at a dose of 1.5-2.0mg/kg (injection time >30 seconds). During induction, the Modified Observer's Assessment of Alertness/Sedation Scale (MOAA/s) score is evaluated every 30±10 seconds; if MOAA/s >1 after 2 minutes, an additional sedative dose (1/2 of the initial dose, injection time ≥10 seconds) is supplemented until MOAA/s ≤1.
  3. Maintenance phase：Continuous intravenous infusion of Propofol Injection at a rate of 4-12mg/kg/h; the dose is adjusted according to Bispectral Index (BIS) to maintain BIS between 40-60. If the patient shows body movement, eye opening, speech or other signs of insufficient se
  Other Names: Dexmedetomidine Injection (nasal spray)
  Arms: Experimental Group ①
Drug: Normal Saline (nasal spray) + Dexmedetomidine Injection (intravenous) + Propofol Injection + Sufentanil Injection — 1. Preoperative intervention：30 minutes before entering the operating room, normal saline is administered via nasal spray in the anesthesia preparation room; 10 minutes before induction, 0.5μg/kg of Dexmedetomidine Injection is given via intravenous injection.
  2. Induction phase：Same as Experimental Group ① (intravenous Sufentanil 0.1μg/kg + Propofol 1.5-2.0mg/kg, with MOAA/s monitoring and supplementary dose rules).
  3. Maintenance phase：Same as Experimental Group ① (continuous Propofol infusion at 4-12mg/kg/h, BIS-adjusted dose, and supplementary sedation rules for insufficient sedation).
  Other Names: Dexmedetomidine Injection (intravenous)
  Arms: Experimental Group ②
Drug: Regular sedation protocol — Preoperative intervention：No dexmedetomidine or normal saline nasal spray; only routine preoperative preparation.
  Induction phase：Same as Experimental Group ① (intravenous Sufentanil 0.1μg/kg + Propofol 1.5-2.0mg/kg, with MOAA/s monitoring and supplementary dose rules).
  Maintenance phase：Same as Experimental Group ① (continuous Propofol infusion at 4-12mg/kg/h, BIS-adjusted dose, and supplementary sedation rules for insufficient sedation).
  Arms: Control Group

SUMMARY:
This prospective randomized single-blind study evaluated the safety and efficacy of combining dexmedetomidine nasal spray with propofol for ERCP (Endoscopic Retrograde Cholangiopancreatography) sedation in eligible patients aged 18-70 years undergoing elective procedures. The primary objectives were to determine: 1) whether this regimen reduced intraoperative hypoxemia (decreased blood oxygen levels), decreased propofol dosage, and improved postoperative recovery quality; 2) to assess nasal administration safety and identify potential medical issues (e.g., abnormal blood pressure or bradycardia) compared to intravenous injection and control group protocols. Participants were randomly assigned to three groups: ① nasal spray group (preoperative nasal spray of dexmedetomidine + propofol), ② intravenous group (preoperative intravenous injection of dexmedetomidine + propofol), ③ and conventional group (propofol alone).

DETAILED DESCRIPTION:
General Information purpose of research：To evaluate the safety and effectiveness of right mebromide nasal spray combined with propofol in endoscopic retrograde cholangiopancreatography.

Patients with no restriction on gender, aged 18-70 years, with a BMI of 18-30 kg/m², and American Society of Anesthesiologists (ASA) physical status Ⅰ or Ⅱ.

Exclusion criteria: - Patients who explicitly refused to participate in the study; - Patients with difficult airway management (modified Mallampati score of Grade IV); - Patients with anemia or thrombocytopenia (Hb < 90 g/L, PLT < 80×10⁹/L); - Patients with abnormal liver or kidney function; - Patients with a history of nasal surgery/trauma or deviated nasal septum; - Patients with allergies or contraindications to dexmedetomidine, opioids, propofol, rocuronium, or their components; - Patients with a history of abnormal recovery from previous surgery or anesthesia.

Patients were divided into three groups using a random number table method: pre-intranasal spray combined with infusion group (PP group), conventional intravenous combined with infusion group (CP group), and control group (C group).

Anesthetic Method All patients fasted from liquids for 4 hours and solids for 8 hours before surgery. Upon entering the pre-anesthesia preparation room, an upper limb venous access was established, and sodium bicarbonate Ringer's solution was infused at a rate of 300 mL/h. After entering the operating room, the patient assumed a "lateral prone position" and received oxygen via a nasal cannula at a flow rate of 5 L/min until the completion of ERCP and full awakening. All ERCP procedures were performed by experienced endoscopists. Non-invasive blood pressure, heart rate, electrocardiogram, pulse oxygen saturation, and bispectral index (BIS) were monitored. An anesthetic machine, laryngeal mask, endotracheal tube, rescue equipment, and drugs were prepared. Anesthetics were infused through the forearm venous access of the patient. Anesthetic induction methods: - Experimental Group ① (PP group): Thirty minutes before entering the operating room, 50-100 μg of dexmedetomidine injection was administered via intranasal spray in the pre-anesthesia preparation room (Administration method: Hold the dexmedetomidine nasal spray upright. Keep the nozzle away from the mouth, nose, eyes, and other body parts. Place the index and middle fingers on both sides of the top of the spray pump, and the thumb at the bottom of the bottle. Press the spray pump downward with uniform force using the index and middle fingers for 7 times, and at least one complete spray should be observed within these 7 presses. Clean the nostrils before use to ensure the nasal cavity is dry and clean. The patient should be in a sitting position with the head slightly tilted forward, and the product should remain upright during use. Insert the nozzle of the nasal spray into the nostril at an angle consistent with the nasal cavity. Press the spray pump downward fully with uniform force using the index and middle fingers (1 spray). After spraying 1 dose into each nostril, tilt the head slightly backward and inhale gently. After a 30-second interval, spray another dose into each nostril, with a total of 2-4 sprays). Upon entering the operating room, induction was performed with intravenous sufentanil (Yichang Renfu Pharmaceutical Co., Ltd.) at a dose of 0.1 μg/kg and propofol (Jiabo Pharmaceutical, Guangdong, China) at a dose of 1.5-2.0 mg/kg (intravenous injection time > 30 seconds). During induction, the modified Observer's Assessment of Alertness/Sedation (MOAA/s) scale score was evaluated every 30±10 seconds. If the MOAA/s score was still > 1 after 2 minutes, additional sedatives were supplemented (supplementary dose = 1/2 of the initial dose, injection time ≥ 10 seconds). When the patient's MOAA/s score ≤ 1, the endoscopist began to insert the endoscope and continued to infuse sedatives. - Experimental Group ② (CP group): Thirty minutes before induction, normal saline was administered via intranasal spray; 10 minutes before induction, 0.5 μg/kg of dexmedetomidine was administered intravenously. Induction was performed with sufentanil (0.1 μg/kg) and propofol (1.5-2.0 mg/kg), and the remaining procedures were the same as those in the PP group. - Control Group (C group): Induction was performed with sufentanil (0.1 μg/kg) and propofol (1.5-2.0 mg/kg), and the remaining procedures were the same as those in the two experimental groups. At the end of ERCP, the MOAA/s score was evaluated every 3 minutes until the patient was fully awake (MOAA/s score = 5 in three consecutive evaluations). After surgery, the Aldrete score was calculated every 5 minutes, and the patient was transferred from the post-anesthesia care unit (PACU) to the ward when the score reached ≥ 9 in three consecutive evaluations.

Management of intraoperative adverse events: - For intraoperative hypoxemia or apnea (SpO₂ < 90% for more than 10 seconds): First, increase the oxygen flow rate by 2 L/min; second, lift the mandible, reduce the depth of anesthesia, and insert a nasopharyngeal airway to improve ventilation. - For intraoperative hypotension (systolic blood pressure < 90 mmHg or mean arterial pressure decreased by 20% relative to baseline for more than 2 minutes): Administer 4-12 μg of norepinephrine intravenously. - For bradycardia (heart rate < 50 bpm for more than 1 minute): Administer 0.3-0.5 mg of atropine intravenously.

Observation Indicators :Primary indicators: Intraoperative hypoxemia (SpO₂ < 90% for more than 10 seconds).Secondary indicators: Circulatory fluctuations: Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR), and pulse oxygen saturation (SpO₂) were recorded at the following time points: on entry to the operating room (T0), after induction (T1), when the endoscope entered the esophagus (T2), during duodenal papillary intubation (T3), when the endoscope was removed (T4), and at awakening (T5). Incidence of intraoperative adverse events: Including cough during endoscope insertion, nausea, vomiting, postoperative agitation, pain score, respiratory depression, and use of vasopressors during surgery. Induction and maintenance dosages of propofol. Evaluation of awakening speed and quality: Extubation time, and Steward score immediately after awakening and 30 minutes after awakening. Assessment of agitation and sedation levels using the Richmond Agitation-Sedation Scale (RSAS); assessment of pain and analgesic requirements within 24 hours after surgery using the Numerical Rating Scale (NRS).

Statistical Analysis Based on the safety evidence of dexmedetomidine and references to previous clinical trials, the incidence of hypoxemia was approximately 13.3% in the dexmedetomidine group and 26.7% in the control group among subjects undergoing elective general anesthesia induction. With a type Ⅰ error rate (α) of 0.05, a type Ⅱ error rate (β) of 0.1, and an attrition rate of 10%, the total sample size (N) was calculated using PASS software to be 180, with N1 = N2 = N3 = 60. Statistical analysis was performed using SPSS 31 software. Measurement data conforming to a normal distribution were expressed as mean ± standard deviation (x±s), and one-way analysis of variance was used for intergroup comparison. Measurement data not conforming to a normal distribution were expressed as median (M) and interquartile range (IQR), and the nonparametric Mann-Whitney U test was used for intergroup comparison. Count data were expressed as cases (%), and the χ² test or Fisher's exact test was used for intergroup comparison. The rank sum test was used for comparison of ordinal data. A P-value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* no restriction on gender,
* aged 18-70 years,
* BMI of 18-30 kg/m²,
* American Society of Anesthesiologists (ASA) physical status Ⅰ or Ⅱ.

Exclusion Criteria:

* Patients who explicitly refused to participate in the study;
* Patients with difficult airway management (modified Mallampati score of Grade IV);
* Patients with anemia or thrombocytopenia (Hb < 90 g/L, PLT < 80×10⁹/L);
* Patients with abnormal liver or kidney function;
* Patients with a history of nasal surgery/trauma or deviated nasal septum;
* Patients with allergies or contraindications to dexmedetomidine, opioids, propofol, rocuronium, or their components;
* Patients with a history of abnormal recovery from previous surgery or anesthesia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2025-10-02 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative hypoxemia | From the start of the surgery to 1 hour after the surgery
  (SpO₂ < 90% for more than 10 seconds)

SECONDARY OUTCOMES:
Blood pressure fluctuations | on entry to the operating room (T0), after induction (T1), when the endoscope entered the esophagus (T2), during duodenal papillary intubation (T3), when the endoscope was removed (T4), and at awakening (T5).
  Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP)
Heart rate fluctuations | on entry to the operating room (T0), after induction (T1), when the endoscope entered the esophagus (T2), during duodenal papillary intubation (T3), when the endoscope was removed (T4), and at awakening (T5).
  heart rate (HR)
SpO₂ fluctuations | on entry to the operating room (T0), after induction (T1), when the endoscope entered the esophagus (T2), during duodenal papillary intubation (T3), when the endoscope was removed (T4), and at awakening (T5).
  pulse oxygen saturation (SpO₂)
Incidence of intraoperative adverse events | From the start of the surgery to 1 hour after the surgery
  Including cough during endoscope insertion, nausea, vomiting, postoperative agitation, pain score, respiratory depression

OTHER OUTCOMES:
dosages of propofol | From the start of the surgery to the end of the surgery
  Induction and maintenance dosages of propofol
Extubation time | From entering the PACU to leaving the PACU
  Extubation time Evaluation of awakening speed and quality
Steward score | From entering the PACU to leaving the PACU
  Steward score immediately after awakening and 30 minutes after awakening. Evaluation of awakening speed and quality
Richmond Agitation-Sedation Scale (RSAS) | From entering the PACU to leaving the PACU
  Assessment of agitation and sedation levels using the Richmond Agitation-Sedation Scale (RSAS). Evaluation of awakening speed and quality
Pain Numerical Rating Scale (NRS) | From entering the PACU to leaving the PACU
  assessment of pain after surgery using the Numerical Rating Scale (NRS).The Numeric Rating Scale (NRS) accurately classifies pain levels using 11 numbers (ranging from 0 to 10), with each number corresponding to a clear pain description. Patients are required to select the number that best matches their current pain based on their own feelings-the higher the number, the more severe the pain. A score of 10 represents the most severe pain, while a score of 0 indicates no pain at all.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyou Wei, PhD, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai East Hospital,Affiliated to Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No